CLINICAL TRIAL: NCT01163344
Title: Dance Exercise as Novel Complementary Therapy for Parkinson's Disease
Acronym: DANCE-PD
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Tarsy, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2010P000029
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Parkinsons Disease
Keywords: Gait, balance, Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dance Therapy Group: This will group will undergo dance therapy once a week for a series of 8 weeks.
- Physical Therapy Group: This group will undergo physical therapy sessions once a week for a series of 8 weeks

SUMMARY:
The purpose of this study is to gather data to see if so-called enriched forms of exercise programs such as dance is more effective in improving balance and quality of life in patients with idiopathic Parkinson's disease than regular exercise programs that are currently provided by physical therapists.

DETAILED DESCRIPTION:
Comparison of traditional PT to dance in people who have parkinsons disease to measure which is better for gait, balance and QOL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD at least 3 years ago
* Less than 80 years of age
* Have gait and balance issues

Exclusion Criteria:

* Diagnosis of PD for less than 3 years
* 80 years of age or older
* Not have gait and balance issues

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To qualify for this study, subject must have been diagnosed with Parkinson's Disease for 3 years or more, be less than 80 years of age, and have problems with gait and balance
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Balance and Gait improvement | 10 weeks
  We seek to determine if balance and gait are improved as a result of dance therapy. This will be compared to the balance and gait data of group physical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tarsy, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Veronique Vanderhorst, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.pdtrials.org